CLINICAL TRIAL: NCT05379725
Title: Mediterranean vs. High-Fermented-Food Diet Adherence on Inflammation and Disease Activity in Systemic Lupus Erythematosus
Brief Title: Mediterranean vs. High-Fermented-Food Diet Adherence on Inflammation in Lupus
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Lack of funding to continue.
Sponsor: University of Florida (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: IRB202200703
Record Dates: First submitted 2022-05-09; First posted 2022-05-18 (Actual); Last update posted 2025-06-26 (Actual); Status verified 2025-06

CONDITIONS: Lupus Erythematosus, Systemic
Keywords: SLE; Lupus; Mediterranean diet; Fermented food; Inflammation
MeSH Terms: conditions — Lupus Erythematosus, Systemic; Inflammation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mediterranean diet (Experimental): Participants will receive diet education on adherence to a Mediterranean dietary pattern.
  Interventions: Other: Mediterranean Dietary Pattern
- Fermented food (Experimental): Participants will receive diet education on adherence to a high fermented food dietary pattern.
  Interventions: Other: High Fermented Food Dietary Pattern

INTERVENTIONS:
Other: Mediterranean Dietary Pattern — The Mediterranean dietary pattern includes whole or minimally processed foods with a high intake of vegetables, fruits, whole grains, fish, and olive oil.
  Arms: Mediterranean diet
Other: High Fermented Food Dietary Pattern — Fermented foods such as yogurt, kefir, fermented cottage cheese, fermented vegetables, vegetable brine drinks, kombucha, other fermented non-alcoholic drinks, and other foods will be recommended.
  Arms: Fermented food

SUMMARY:
This is a 4-month randomized controlled trial to evaluate the feasibility of 'good and very good' adherence to the Mediterranean dietary pattern and to a high-fermented-food diet by individuals with Systemic lupus erythematosus (SLE).

DETAILED DESCRIPTION:
Given the demonstrated beneficial effects of the Mediterranean dietary pattern in autoimmune disease and the potential benefit of a high-fermented-food diet on inflammatory profiles, we aim to determine the feasibility and relative benefit of a Mediterranean dietary pattern versus a high-fermented-food diet on inflammatory markers and clinical outcomes in individuals with SLE. The primary aim of the study is to evaluate the feasibility of 'good and very good' adherence to the Mediterranean dietary pattern and to a high-fermented-food diet by individuals with SLE. Secondary aims will determine the effects of the Mediterranean dietary pattern and a high-fermented-food diet on attenuating inflammation and disease activity in individuals with SLE. This is a 4-month randomized controlled trial with a 1-month baseline of usual diet and 3-month intervention. Participants will complete the online DHQ III and diet adherence questionnaires monthly. Blood will be obtained at randomization and at the end of the intervention period for analysis of inflammatory cytokines. Dietary intake during baseline and intervention will be assessed by 5, ASA 24-h dietary recalls.

ELIGIBILITY:
Inclusion Criteria:

* > 18 years of age
* Able to provide informed consent and undertake study questionnaire completion in English
* Meets SLE diagnostic criteria and is currently under the care of a rheumatologist, nephrologist, or other physician regarding SLE care
* Be willing and able to comply with all the study-related procedures

Exclusion Criteria:

* Pregnant or planning pregnancy within the duration of the interventional study.
* Currently following a vegetarian/vegan diet.
* Allergy/sensitivity to gluten, soy, or cow's milk.
* Self-disclosure of lactose intolerance
* Inability to comply with the study procedures.
* Baseline dietary fiber intake > 30 g/day
* MEDAS score at baseline > 9
* Baseline consumption of > 2 servings per day of fermented foods

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2022-03-22 (Actual); Primary Completion 2025-03-01 (Actual); Study Completion 2025-03-01 (Actual)

PRIMARY OUTCOMES:
Adherence - Mediterranean Diet | baseline, month 1, 2 and 3
  Percent of participants achieving 'good to very good adherence') as assessed by the 14-day Mediterranean diet questionnaire (MEDAS) score
Adherence - Fermented Food Diet | baseline, month 1, 2, and 3
  Percent of participants achieving > 5 servings of fermented foods per day

SECONDARY OUTCOMES:
Diet Quality | baseline, month 3
  Healthy Eating Index 2015 score (0 minimum to 100 maximum). Higher values indicate better diet quality.
Systemic Lupus Erythematosus Disease Activity | baseline, month 3
  Systemic Lupus Erythematosus disease activity using the Systemic Lupus Erythematosus Disease Activity Index 2000 (SLEDAI-2K) score (0 minimum and 105 maximum, with higher scores representing higher disease activity.
ESR | baseline, month 3
  Erythrocyte sedimentation rate
hsCRP | baseline, month 3
  high-sensitivity C-reactive protein
anti-dsDNA | baseline, month 3
  Anti-double stranded DNA
Cytokine profile | baseline, month 3
  Cytokines profile e.g., interleukin-18 (IL-18), tumor necrosis factor (TNF), IL-6, IL-2, IL-10

CONTACTS AND LOCATIONS:
Locations (1):
- University of Florida/UF Health, Gainesville, Florida, United States

IPD SHARING:
Plan to Share IPD: No